CLINICAL TRIAL: NCT07187570
Title: RECURrence of Atrial Fibrillation After Cardioversion of Patients Randomized to Open-label Treatment With Dapagliflozin or Usual Care
Brief Title: RECURrence of Atrial Fibrillation After Cardioversion of Patients Randomized to Dapagliflozin or Usual Care
Acronym: RECUR-AF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EU CT 2024-513719-28-00; 2024-513719-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-03; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation (AF)
Keywords: dapagliflozin; sodium-glucose transport-2 inhibitor; electric cardioversion; hand-held ECG device
MeSH Terms: conditions — Atrial Fibrillation | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Prospective randomized open blinded end-point (PROBE) study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Standard of care
- Dapagliflozin (Experimental): Tablet Dapagliflozin 10 mg once daily
  Interventions: Drug: Dapagliflozin 10 mg once daily

INTERVENTIONS:
Drug: Dapagliflozin 10 mg once daily — Tablet Dapagliflozin 10 mg orally during from randomization for maximum 56 days.
  Arms: Dapagliflozin

SUMMARY:
The goal of this clinical trial is to learn if drug dapagliflozin, a sodium-glucose transport-2 inhibitor, works to treat atrial fibrillation in adults. The main question it aims to answer is:

• Does the drug dapagliflozin reduce the recurrence rate of atrial fibrillation?

Researchers will compare drug dapagliflozin to standard therapy to see if drug dapagliflozin reduce the recurrence of atrial fibrillation.

Persons with atrial fibrillation who are planned for an electric cardioversion will:

* Take the drug dapagliflozin, or no drug, once a day for a maximum of 56 days
* Undergo a planned electric cardioversion of the atrial fibrillation
* Record the rhythm with a hand-held device that transmits the signal to researchers during the study period, but no longer than for 56 days

ELIGIBILITY:
Inclusion Criteria:

* Patients with AF on ECG who are planned for electrical cardioversion within 7-26 days from inclusion-date.
* Age ≥ 55 years.
* Provided written informed consent.

Exclusion Criteria:

* Current treatment with an SGLT2 inhibitor.
* Prior/current diagnosis of heart failure.
* Type 1 diabetes mellitus.
* Estimated glomerular filtration rate (eGFR) < 25 mL/min/1.73m2.
* Pulmonary vein isolation within preceding 3 months or planned pulmonary vein isolation during the study period (56 days).
* Contraindications to SGLT2 inhibitors.
* Any condition or circumstance in which the patient should not participate in the study according to the study investigator.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence | 30 days after elective electrical cardioversion
  Time to first AF recurrence detected with an ECG- monitoring device within 30 days after planned elective electrical cardioversion.

SECONDARY OUTCOMES:
Proportion of patients in SR at 30 days | 30 days after elective electrical cardioversion
  Proportion of patients in SR 30 days after cardioversion.
Proportion of patients without any atrial fibrillation recurrence at 30 days | 30 days after elective electrical cardioversion
  Proportion of patients without any atrial fibrillation recurrence at 30 days
Time to spontaneous return to sinus rhythm before electrical cardioversion | Up to 26 days
  Time to spontaneous return to sinus rhythm measured from randomization to electrical cardioversion (max 26 days)
Spontaneous return to sinus rhythm before cardioversion. | Up to 26 days
  Number of patients with return to sinus rhythm at time of electrical cardioversion (maximum 26 days from randomization)
Success of cardioversion | Periprocedural
  Discharged with sinus rhythm after electric cardioversion
Total number of days with atrial fibrillation | From day of electric cardioversion to 30 days after
  Total number of days with AF recordings during the 30 days following cardioversion.
Absence of clinical atrial fibrillation recording | From randomization to 30 days after electric cardioversion
  Absence of clinical atrial fibrillation recurrence (12-lead ECG-verified) during follow-up after cardioversion or after spontaneous return to SR (before cardioversion).

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Szummer, MD PhD, Principal Investigator — Karolinska Institutet; Ziad Hijazi, MD PhD, Principal Investigator — Dept. of Medical Sciences, Uppsala University, Uppsala, Sweden
Locations (7):
- Sweden (7):
  - Linköping university hosptial, Linköping
  - Örebro University hospital, Örebro
  - Södersjukhuset, Stockholm
  - Karolinska University Hospital, Stockholm
  - Danderyds Hospital, Stockholm
  - Norrlands universitetssjukhus, Umeå
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: No